CLINICAL TRIAL: NCT05712889
Title: An Open-label, Multicenter Phase 1 Study to Characterize Safety, Tolerability, Preliminary Antitumor Activity and Pharmacokinetics of VIP236 Monotherapy in Subjects With Advanced Cancer
Brief Title: Phase 1 Dose Escalation Study for VIP236 in Patients With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vincerx Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: VNC-236-101
Record Dates: First submitted 2023-01-25; First posted 2023-02-06 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Neoplasms
Keywords: VIP236; Solid tumors; Biliary tract cancer; Breast cancer; Small cell lung cancer; Triple negative breast cancer; Cervical cancer; Gastric cancer; Lung cancer; Non-small cell lung cancer; Ovarian cancer; Pancreatic adenocarcinoma; Advanced solid tumors; Metastatic cancer; Endometrial cancer; Urothelial cancer
MeSH Terms: conditions — Neoplasms; Biliary Tract Neoplasms; Breast Neoplasms; Small Cell Lung Carcinoma; Triple Negative Breast Neoplasms; Uterine Cervical Neoplasms; Stomach Neoplasms; Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Ovarian Neoplasms; Neoplasm Metastasis; Endometrial Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Escalation of VIP236 (Q3W) (Experimental): Investigating VIP236 in a dose escalation cohort in subjects with advanced solid tumor cancer. Dosing occurs on D1 of each 21-day cycle
  Interventions: Drug: VIP236 (Q3W)
- Dose Escalation of VIP236 (Q2W) (Experimental): Investigating VIP236 in a dose escalation cohort in subjects with advanced solid tumor cancer. Dosing occurs on D1 and D15 of each 28-day cycle.
  Interventions: Drug: VIP236 (Q2W)

INTERVENTIONS:
Drug: VIP236 (Q3W) — VIP236 will be administered by IV infusion once every 3 weeks, for a 21-day cycle.
  Arms: Dose Escalation of VIP236 (Q3W)
Drug: VIP236 (Q2W) — VIP236 will be administered by IV infusion once every 2 weeks, for a 28-day cycle.
  Arms: Dose Escalation of VIP236 (Q2W)

SUMMARY:
Determine the safety, tolerability, and maximum tolerated dose (MTD) of IV administered VIP236 as monotherapy in patients with advanced solid tumor cancer

DETAILED DESCRIPTION:
Solid tumor subjects with histologically confirmed advanced or metastatic disease who have relapsed or refractory to standard of care. Subjects must have exhausted all available standard therapies or be deemed ineligible for potential available therapies.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged >/=18 years, able to provide informed consent and willing to comply with all study procedures.
* Histologically confirmed advanced or metastatic solid tumors that are relapsed or refractory to standard of care. Subjects must have exhausted all available standard therapies or be deemed ineligible for potential available therapies. Refer to NCCN guidelines of each respective histology for guidance. Starting with Amendment 3, this study will focus enrollment on the following cancers:

Biliary tract cancers Breast cancer Cervical cancer Endometrial carcinoma Gastric cancer/gastroesophageal junction adenocarcinoma Nonsmall cell lung cancer Ovarian cancer/fallopian tube cancer/primary peritoneal cancer Pancreatic adenocarcinoma Small cell lung cancer Urothelial cancer

* Adequate bone marrow, liver, and renal functions.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.

Exclusion Criteria:

* Subjects who have new or progressive brain or meningeal or spinal metastases.
* Clinically significant cardiac disease including congestive heart failure > New York Heart Association (NYHA) Class II), evidence for coronary artery disease (eg, unstable angina (anginal symptoms at rest) or new-onset angina (within the last 6 months or myocardial infarction within the past 6 months before first dose.
* Major surgery or significant trauma within 4 weeks before the first dose of study drug.
* Medical history of chronic obstructive pulmonary disease (COPD) and other respiratory disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2023-01-24 (Actual); Primary Completion 2024-10-10 (Actual); Study Completion 2024-10-10 (Actual)

PRIMARY OUTCOMES:
Incidence of DLT (Dose limit toxicity) of VIP236 | Cycle 1 Day 1 through Cycle 2 Day 1, where each cycle is up to 28 days
Number of participants with adverse events as a measure safety and tolerability | Cycle 1 Day 1 up to 30 days after the last dose, where each cycle is up to 28 days (up to approximately 10 months)

SECONDARY OUTCOMES:
Objective response rate (ORR), defined as the proportions of subjects who have a best overall response of partial response (PR) or complete response (CR) as determined by investigators using RECIST 1.1 | Up to 24 onths
Disease control rate (DCR) per RECIST v1.1, defined as best overall response of complete response (CR), partial response (PR), or stable disease (SD) as determined by Investigator review. | Cycle 1 Day 1 up to 30 days after the last dose, where each cycle is up to 28 days (up to approximately 10 months)
Progression-free survival per RECIST v1.1, defined as the time from enrollment to documented disease progression or death from any cause, whichever occurs earlier as determined by Investigator review | Up to 24 months
Maximum observed drug concentration in measured matrix after single dose administration (Cmax) of VIP236 | Cycle 1 Day 1 through Cycle 2 Day 1, where each cycle is up to 28 days
Area under the concentration versus time curve from zero to infinity after single (first) dose (AUC) of VIP236 | Cycle 1 Day 1 through Cycle 2 Day 1, where each cycle is up to 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Vincerx Study Director, Study Director — Vincerx Pharma, Inc.
Locations (6):
- United States (3):
  - Honor Health, Scottsdale, Arizona
  - NEXT Austin, Austin, Texas
  - NEXT Oncology San Antonio, San Antonio, Texas
- Australia (3):
  - Macquarie University, Macquarie Park, New South Wales
  - ICON Brisbane, Brisbane, Queensland
  - ICON Adelaide, Adelaide, Southern Australia